CLINICAL TRIAL: NCT02243241
Title: A Randomized, Double-blind, Placebo- and Positive-Controlled, Parallel Group, Dose Escalating Study of the Effect of Hydrocodone Bitartrate (HYD) Extended-Release Tablets at Doses up to 160 mg on QT/QTc in Healthy Adult Subjects
Brief Title: The Effect of Hydrocodone Bitartrate (HYD) Extended-Release Tablets on QT /QTc Intervals in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: HYD1009
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Healthy volunteers; Opioid; ECG; QTcI
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- HYD (Experimental)
  Interventions: Drug: HYD; Drug: Placebo for moxifloxacin
- Moxifloxacin (Other): Moxifloxacin is the positive control.
  Interventions: Drug: Moxifloxacin; Drug: Placebo for HYD
- Placebo (Placebo Comparator): Placebo for HYD and placebo for moxifloxacin
  Interventions: Drug: Placebo for HYD; Drug: Placebo for moxifloxacin

INTERVENTIONS:
Drug: HYD — Hydrocodone bitartrate 80 mg (day 9), 120 mg (day 12), 160 mg [(1) 40 mg tablet + (1) 120 mg tablet] (day 15) extended-release tablets administered orally every 24 hours.
  Arms: HYD
Drug: Moxifloxacin — Moxifloxacin 400 mg tablets administered orally on the morning of day 9, day 12, and day 15 only.
  Other Names: Avelox®
  Arms: Moxifloxacin
Drug: Placebo for HYD — Placebo to match HYD tablets administered orally every 24 hours.
  Arms: Moxifloxacin; Placebo
Drug: Placebo for moxifloxacin — Placebo to match moxifloxacin tablets administered orally on the mornings of day 9, day 12, and day 15 only.
  Arms: HYD; Placebo

SUMMARY:
Evaluate the effect of multiple doses (once daily for 3 days each of HYD 80, 120, and 160 mg tablets) on the QT/QTc interval.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent;
* Body weight ranging from 50 to 100 kilograms (kg) [110 to 220 pounds] and body mass index (BMI) of 18 to 30 (kg/m2);
* Males and females aged 18 to 50 years;
* Willing to eat the food supplied during the study;
* Willing to refrain from strenuous exercise through the end-of-study visit. Subjects did not begin a new exercise program nor participate in any unusually strenuous physical exertion;
* Healthy and free of significant abnormal findings as determined by medical history, physical examination, clinical laboratory values, vital signs, and safety 12-lead ECG;
* Females of childbearing potential must use an adequate and reliable method of contraception (ie, barrier with additional spermicidal foam or jelly, intra-uterine device, hormonal contraception). Females who are postmenopausal must be postmenopausal for ≥ 1 year and have elevated serum follicle stimulating hormone (FSH).

Exclusion Criteria:

* Females who are pregnant (positive beta human chorionic gonadotropin test) or lactating;
* Current or recent (within 5 years) history of drug or alcohol abuse;
* History or any current conditions that may interfere with drug absorption, distribution, metabolism, or excretion;
* Use of an opioid-containing medication in the past 30 days preceding the initial dose in this study;
* Known allergy to hydrocodone, opioids, psychotropic or hypnotic drugs, moxifloxacin, or any member of the quinolone class drugs;
* Any history of frequent nausea or emesis regardless of etiology;
* Any history of seizures or head trauma with sequelae;
* Participation in a clinical drug study during the 30 days preceding the initial dose of study drug in this study;
* Use of any medication including thyroid hormonal therapy (hormonal contraception and hormonal replacement therapy in the form of estrogen with or without progestin is allowed), vitamins, herbal and/or mineral supplements during the 7 days preceding the initial dose of study drug;
* Any significant illness during the 30 days preceding the initial dose of study drug in this study;
* Any personal or family history of prolonged QT interval or disorders of cardiac rhythm;
* Abnormal cardiac conditions including hypertension;
* Abnormal cardiac condition denoted by any of the following:

  * QT data corrected for heart rate using the Fridericia formula (QTcF) interval >450 milliseconds (msec)
  * PR interval >240 msec or QRS >110 msec
  * Evidence of second- or third-degree atrioventricular block
  * Pathological Q-waves (defined as Q-wave >40 msec or depth >0.5 millivolts [mV])
  * Evidence of ventricular pre-excitation, complete left bundle branch block (LBBB), right bundle branch block (RBBB), or incomplete RBBB
  * With a resting heart rate (HR) outside the range of 40 to 90 beats per minute (bpm);
* Abnormalities on physical examination, vital signs, safety 12-lead ECG, or clinical laboratory values, unless those abnormalities are judged clinically insignificant by the investigator;
* Oxygen saturation <94% as measured by pulse oximetry (SpO2);
* Refusal to abstain completely from caffeine or xanthine during confinement;
* Refusal to abstain from consumption of alcoholic beverages 48 hours prior to initial study drug administration through the end-of-study visit;
* Blood or blood products donated within 30 days prior to initial study drug administration or any time through the end-of-study visit, except as required by the study protocol;
* History of smoking or use of nicotine products within 45 days of initial study drug administration or a positive urine cotinine test;
* Positive results of urine drug screen or alcohol screen;
* Positive results of hepatitis B surface antigen (HBsAg), hepatitis C antibody (anti-HCV);
* Presence of Gilbert's Syndrome or any known hepatobiliary abnormalities;
* The investigator believes the subject to be unsuitable for reason(s) not specifically stated in the exclusion criteria.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The time-matched analysis on QT data (change from baseline, placebo-subtracted) corrected for heart rate (QTc), based on an individual correction (QTcI) method | Baseline and Day 9
  The electrocardiogram (ECG) effects of HYD 80 mg (day 9) on the QT/QTc interval
The time-matched analysis on QT data (change from baseline, placebo-subtracted) corrected for heart rate (QTc), based on an individual correction (QTcI) method | Baseline and Day 12
  The ECG effects of HYD 120 mg (day 12) on the QT/QTc interval
The time-matched analysis on QT data (change from baseline, placebo-subtracted) corrected for heart rate (QTc), based on an individual correction (QTcI) method | Baseline and Day 15
  The ECG effects of HYD 160 mg (day 15) on the QT/QTc interval

SECONDARY OUTCOMES:
The time-matched analysis on QT data (change from baseline, placebo-subtracted) corrected for heart rate (QTc), based on an individual correction (QTcI) method | Baseline and Day 9
  The ECG effects of moxifloxacin (day 9) on the QT/QTc interval
The time-matched analysis on QT data (change from baseline, placebo-subtracted) corrected for heart rate (QTc), based on an individual correction (QTcI) method | Baseline and Day 12
  The ECG effects of moxifloxacin (day 12) on the QT/QTc interval
The time-matched analysis on QT data (change from baseline, placebo-subtracted) corrected for heart rate (QTc), based on an individual correction (QTcI) method | Baseline and Day 15
  The ECG effects of moxifloxacin (day 15) on the QT/QTc interval

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States